CLINICAL TRIAL: NCT06656208
Title: Effects of Pubic Symphysis Manipulation in Patients With Sacroiliac Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIUMalihaFatima
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: Sacroiliac joint dysfunction; Symphysis pubis dysfunction (SPD); Pubic symphysis manipulation (PSM); Low back pain; Disability; Pubic malalignment
MeSH Terms: conditions — Pelvic Girdle Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Pubic symphysis manipulation with 5 repetitions hold for 10 sec and ask the patient to apply max. Contraction and then relax. Whereas, the therapist applies a rapid stretch to a new barrier and is held for 10 seconds.
  SIJ mobilizations will be given with 30 Oscillations per set for 15 seconds, 3 sets on effected side along with
  Interventions: Other: Pubic symphysis manipulation
- Control Group (Active Comparator): SIJ mobilizations will be given with 30 Oscillations per set for 15 seconds, 3 sets on effected side.
  Interventions: Other: Traditional sacroiliac treatment

INTERVENTIONS:
Other: Pubic symphysis manipulation — Manipulation was applied in the crook lying position with 5 repetitions hold for 10 sec and ask the patient to apply max. Contraction in Abduction and then relax. Whereas, the therapist applies a rapid stretch to a new barrier and is held for 10 seconds.
  Arms: Experimental Group
Other: Traditional sacroiliac treatment — Mobilization was applied in prone lying position on sacroiliac joint, 30 Oscillations per set for 15 seconds, 3 sets on effected side.
  Arms: Control Group

SUMMARY:
The aim of this research is to determine the effect of Pubic Symphysis manipulation on pain, disability and fear avoidance behavior in patients with sacroiliac joint dysfunction. Randomized controlled trials was done at Pakistan Railway Hospital. The sample size was 44. The subjects will be divided into Control group and Experimental group. Each group will be having 22 participants. Study duration was of 12 months. Sampling technique applied was non probability connivance sampling technique. Subject included in the study will be female with presence of back pain for ≥6 months, Unilateral back pain, Age 25-60 years, Postpartum women, Patient with pubic tenderness. Tools used in the study are NPRS, Oswestry Disability Index and FABQ. Data will be analyzed using SPSS version 26.

DETAILED DESCRIPTION:
Sacroiliac joint (SIJ) dysfunction is a degenerative condition that is considered a major cause of low back pain. It has been resulting from abnormal motion of the joint known as SIJ dysfunction (SIJD). During pregnancy, heightened levels of estrogen and relaxin, coupled with the pressure exerted by a growing fetus, may induce excessive mobility in the SIJs. Conversely, pelvic fractures and a sedentary lifestyle can contribute to decreased mobility and fixation of the joints. Life time prevalence of low back pain is 85%. Among these patients 10% to 25% of, sacroiliac joint is the cause of pain. In Pakistan, female undergraduate students have a higher prevalence of low back pain compared to males. Individuals with SIJD often present with unilateral pain below L5. The pain is often localized distal and medial to the PSIS. It is described as sharp, dull, or shooting and is often misdiagnosed as radicular pain, as it can extend down the posterior thigh to the S1 dermatome. Factors contributing to SIJD include high velocity trauma, degenerative arthritis, inflammatory arthropathy etc. The ability to rise from a chair is a basic functional task that is frequently compromised in individuals diagnosed with SIJD. This condition has been associated with up to 14-20% of patients affected by limiting the overall quality of life.

The pubic symphysis plays a vital role in stabilizing the anterior pelvis while allowing for a limited range of movement. Pubic symphysis dysfunction is characterized by discomfort in the pubic bone region that intensifies during activities such as walking, lifting, or stair climbing, hip abduction, rolling over in bed. Patients often report tenderness over the pubic symphysis. Symptoms include burning, stabbing, or shooting pain that radiates towards the abdomen, back, leg, and perineum. Symphysis pubis dysfunction (SPD) occurs where the joint becomes sufficiently relaxed to allow instability in the pelvic girdle. In severe cases of SPD the symphysis pubis may partially or completely rupture.

Literature review: A study by Aghalar Javadov et al. in 2021 aims to assess the effects of manual therapy for sacroiliac joints in comparison with lumbar exercises. Result of this study shows long term effects of manual therapy in sacroiliac joint dysfunction.

Another study conducted by Shokri E et al. in which effectiveness of sacroiliac joint (SIJ) manipulation alone was compared with a combination of SIJ and lumbar manipulation for treating SIJ dysfunction. The study results indicated that a single session of SIJ and lumbar manipulation is more effective in reducing functional disability compared to SIJ manipulation alone.

A study conducted by S. Becker et al. investigates whether sacroiliac joint pain is linked to alterations in the pubic symphysis. The findings of this study indicate that changes in the pubic symphysis, along with low back pain and positive provocative tests, could potentially indicate dysfunction in the sacroiliac joint.

Purpose of the study was to investigate effects of pubic symphysis manipulation in patients with sacroiliac joint dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age 25-60 years
* Presence of back pain for ≥6 months
* Postpartum women
* Patient with pubic tenderness
* Patient with pubic symphysis asymmetry
* Unilateral back pain
* Participants had 2 positive test out of four test, Sacroiliac distraction test, Sacroiliac compression test, thigh thrust test, sacral thrust test.

Exclusion Criteria:

* Participants underwent surgical approaches
* History of fracture
* Patients suffering from pubic neuralgia and osteitis pubis
* SIJ or Hip joint pathology
* Arthritides
* Adductor strain

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female are prone to SIJ Dysfunction than male, due to pregnancy, joint pain and obesity
Enrollment: 44 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | baseline to 6th day
  The NPRS is a self-reported, or clinician administered, measurement tool to measure pain intensity consisting of a numerical point scale with extreme anchors of 'no pain' to 'extreme pain'. The scale is typically set up on a horizontal or vertical line, ranges most commonly from 0-10 or 0-100, and can be administered in written or verbal form.
Fear Avoidance Belief Questionnaire (FABQ) | baseline to 6th day
  his scale is used to measure fear avoidance behavior in patients due to pain. It consists of 16 items and patients rate their agreement with each statement on a 7- point Likert scale (0 = completely disagree, 6 = completely agree). The original factor analysis revealed two sub-scales: the work sub-scale (FABQ w) with 7 questions (maximum score = 42) and the physical activity sub-scale (FABQ pa) with 4 questions (maximum score = 24). A higher score indicates more strongly held fear avoidance beliefs.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | baseline to 6th day
  The Oswestry Disability Index is used to measure a patient's permanent functional disability. There are 10 questions, for each question there is a possible 5 points; 0 for the first answer, 1 for the second answer, etc. Add up the total for the 10 questions and rate them on the scale at right. Indicating Mild, Moderate, Severe, Complete or No disability.

CONTACTS AND LOCATIONS:
Overall Officials: Maliha Fatima, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No